CLINICAL TRIAL: NCT03269305
Title: An Audit on Management of Chronic Diarrhea
Acronym: AAOMOCD
Status: Completed | Type: Observational
Sponsor: Gehad Adel Mohammed (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Gehad Adel Mohammed, principal investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: AssiutU71515
Record Dates: First submitted 2017-08-22; First posted 2017-08-31 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-11

CONDITIONS: Chronic Diarrhea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is to assess whether the staff in gastroenterology unit are sticking to the agreed up on unit's protocol in management of chronic diarrhea over the period of one year(september 2017-september 2018)

DETAILED DESCRIPTION:
chronic diarrhea is defined as having loose or watery stools more than three times aday.Awakening at night to pass stools us often sign of an organic cause of diarrhea.In some cases chronic diarrhea is the result of intestinal infection that persists longer than expected. In other cases chronic diarrhea is apart of a systemic illness.

Etiology:

1. post enteritis diarrhea syndrome in whic small intestinal mucosal damage persists after acute gastroenteritis.Also secondary disaccharidase deficiency and reinfection may be a cause.
2. infectious causes:enteric infection is an important cause.Associated conditions may be T.B or impaired immunity as in malnutrition potentiating the likely-hood of prolonging or acquiring another infection.Viral infection like Rota virus,parasites as E.coli,Giardia lamblia as well as amebiasis have been implicated in chronic diarrhea.
3. Cytomegalovirus on the other hand may act as an opportunistic agent in immuno compromised patients.
4. Non infectious causes include cow's milk allergy,lactose intolerance and inflammatory bowel disease,all of which may cause chronic diarrhea that is often associated with abdominal pain with or without elevated levels of inflammatory markers.
5. Malabsorption syndrome e.g Celiac disease,cystic fibrosis where the stools are usually fatty in nature and bulky in amount.

Good management of chronic diarrhea must include investigations and treatment.A protocol must be followed accurately therefore.

Methodology:

measurment of the degree of sticking of staff in Gastro-enterology unit to the agreed upon unit's protocol in management of chronic diarrhea over the period of one year (September 2017-September 2018).

ELIGIBILITY:
Inclusion Criteria:

* age group from 2 months to 18 years
* cases with diarrhea lasts 2 weeks or more
* Genetically free

Exclusion Criteria:

* age group from 0-2 months
* age group above 18 years
* cases with diarrhea less than 2 weeks
* Gentic disease

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: an audit
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
proper management of chronic diarrhea | september 2017-september 2018
  start accurate treatment of chronic diarrhea by reaching a definitive cause of each case .
  decrease the incidence of undiagnosed cases of chronic diarrhea

CONTACTS AND LOCATIONS:
Overall Officials: Faisal Alkhateeb, Phd, Study Director — Assiut University
Locations (1):
- Gehad, Asyut, Egypt